CLINICAL TRIAL: NCT07002762
Title: Multicentre, Double-blind, Randomized, Placebo-controlled Trial of Clinical Efficacy of Burdock Root Extract in Patients With Asymptomatic Hyperuricaemia
Brief Title: Clinical Efficacy Trial of Burdock Root Extract in Patients With Asymptomatic Hyperuricaemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OMNIFARMA LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Аrctilappa-100-25
Record Dates: First submitted 2025-04-14; First posted 2025-06-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hyperuricemia or Gout
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burdock ( Arctium lappa L.) root extract in a form of a nutritional additive. (Active Comparator): Gastric soluble capsules each containing: 750 mg of burdock ( Arctium lappa L.) root extract in the form of a nutritional additive. The investigational product is packed in identical plastic containers marked as "Investigational Medicinal Product."
  Interventions: Dietary Supplement: Burdock ( Arctium lappa L.) root extract in a form of a nutritional additive; Other: Placebo
- Placebo (Placebo Comparator): Gastric soluble capsules each containing: Maltodextrin, silicon dioxide, calcium stearate, food colourants. The placebo is packed in identical plastic containers marked as "Placebo."
  Interventions: Dietary Supplement: Burdock ( Arctium lappa L.) root extract in a form of a nutritional additive; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Burdock ( Arctium lappa L.) root extract in a form of a nutritional additive — Gastric soluble capsules each containing: 750 mg of burdock ( Arctium lappa L.) root extract in the form of a nutritional additive
  Other Names: LOPUNID; URICA-EURIKA
Other: Placebo — Gastric soluble capsules each containing: Maltodextrin, silicon dioxide, calcium stearate, food colourants

SUMMARY:
Multicentre, double-blind, randomized, placebo-controlled trial of the clinical efficacy of burdock root extract in patients with asymptomatic hyperuricemia, with the primary objective to assess the efficacy of the use of burdock root extract in patients with asymptomatic hyperuricaemia versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricaemia confirmed by a laboratory, uric acid level from 360 to 540 μmol/L in women and from 420 to 540 μmol/L in men;

  * Age from 35 to 65 years at the baseline;
  * Patients examined by an experienced specialist not revealing any clinical evidences of gout or other somatic consequences of hyperuricaemia;
  * Not taking any other nutritional additives;
  * Women of reproductive age having negative pregnancy test at the baseline and at the end of the trial;
  * Not taking any diuretics, or their administration based on a regimen usual for a patient, without changes;
  * Not taking part in any other clinical trials;
  * Consent and voluntarily signed informed consent form for participation in the clinical trial.

Exclusion Criteria:

* Age <35 or >65 years;
* Fever (above 36.8 оС);
* Pregnancy and lactation;
* Patients with any somatic evidences of hyperuricaemia including gout taking antigout drugs during or within 6 months before the trial;
* Patients with mental disorders / taking antipsychotics or antidepressants;
* Patients not giving (informed) consent to participate in the trial;
* Patients causing doubts of the study doctor as to their motivation to comply with the trial;
* Presence of any concomitant decompensated diseases or acute conditions able to influence results of the trial;
* Alcohol abuse and drug addiction;
* Changes in taking diuretics within a month before and during the trial;
* Participation in any other clinical trial;
* Taking any nutritional additives.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Body temperature | 0 - 60 days
Body weight | 0 - 60 days
  kg
Body mass index | 0 - 60 days
Purpouse of the trial | Till end of 2025 year
  1. To study blood levels of uric acid before and after the two-months administration of IMP and placebo in a dose of 1 capsule twice per day in patients with asymptomatic hyperuricaemia and a baseline level of uric acid from 360 to 540 μmol/L in women and from 420 to 540 μmol/L in men.
  2. To study safety of administration of IMP.

SECONDARY OUTCOMES:
Uric acid | 0 - 60 days
  μmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- State Institution "National Research Centre "Academician M. D. Strazhesko Institute of Cardiology, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided